CLINICAL TRIAL: NCT06984575
Title: Relationship Between Intestinal Flora Changes and Hyperuricemia Under Chronic Psychological Stress
Status: Completed | Type: Observational
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Zhang Manna, Director, Principal Investigator, Clinical Professor, Shanghai 10th People's Hospital
Other Study IDs: stress and hyperuricemia
Record Dates: First submitted 2024-02-21; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Hyperuricemia
MeSH Terms: conditions — Hyperuricemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum Sample Collection# and Stool specimen collection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- LSC: healthy people with low level of stress
  Interventions: Other: No interventions
- HSC: healthy people with high level of stress
  Interventions: Other: No interventions
- LSH: hyperuricemia patients with low level of stress
  Interventions: Other: No interventions
- HSH: hyperuricemia patients with high level of stress
  Interventions: Other: No interventions

INTERVENTIONS:
Other: No interventions — No interventions

SUMMARY:
To clarify the mechanism of stress on the incidence of hyperuricemia

DETAILED DESCRIPTION:
To clarify the differences in intestinal microorganisms and metabolism between healthy people and hyperuricemia patients and across different level of stress

ELIGIBILITY:
Inclusion Criteria:

1. Obtain the informed consent of the subjects before conducting any trial-related activities;
2. Males aged 18-69;
3. The hyperurcemia group must meet the diagnostic criteria of having blood uric acid >420umol/L measured twice on an empty stomach on different days under a normal purine diet;

Exclusion Criteria:

- 1)Use of any uric acid-lowering drugs, anti-gout drugs, steroids, proton pump inhibitors, or non-steroidal anti-inflammatory drugs within one month before enrollment; 2)Use of any antibiotics, probiotics, or other drugs including traditional Chinese medicine within one month before enrollment; 3)Abnormal liver function, ALT and AST are more than 2.5 times the upper limit of normal; 4)Other diseases that affect glucose and lipid metabolism: hyperthyroidism, hypothyroidism, hypercortisolism, etc.

5)Chronic kidney disease or severe renal impairment, according to eGFR grading <45mL/min/1.73m2; 6)Secondary hyperuricemia 7)Any gastrointestinal diseases

Ages: 18 Years to 69 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hyperuricemia patients and healthy controls
Sampling Method: Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Phenotype differences in the gut microbiome by metagenomic sequencing. | Samples to be collected once per participant within 7 days of enrollment
  including microbial composition analysis(Taxonomic Annotation Tools: MetaPhlAn4; Functional Gene Analysis Tools:eggNOG-mapper (functional classification) and diversity metrics(α-diversity (Shannon index) and β-diversity (Bray-Curtis distance, UniFrac distance)
sequencing results of the fecal metabolome in the population | Samples to be collected once per participant within 7 days of enrollment

SECONDARY OUTCOMES:
Serum uric acid | Samples to be collected once per participant within 7 days of enrollment
  Uric acid in umol/L.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Tenth People's hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided